CLINICAL TRIAL: NCT00932867
Title: Surveillance of Efficacy and Safety of Drug PRITOR in patieNts With Arterial Hypertension, Who do Not Tolerate ACE inhibitoR Treatment
Acronym: SONAR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer spol.s.r.o.
Other Study IDs: 14010; 14010 - KL0711SK; 14327 - KL0711RO
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension
Keywords: Arterial Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Kinzal/Pritor (Telmisartan, BAY68-9291)

INTERVENTIONS:
Drug: Kinzal/Pritor (Telmisartan, BAY68-9291) — Patients under daily life treatment receiving Pritor according to local drug information.

SUMMARY:
Surveillance of efficacy and safety of drug PRITOR in patieNts with arterial hypertension, who do not tolerate ACE inhibitoR treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Arterial hypertension (SBP < 160 mmHg and DBP < 100 mmHg)
* Patients, who do not tolerate ACE inhibitors (must be documented in the official ambulant documentation)

Inclusion criteria for the control arm (treated by ACEi):

* Patients over 18 years of age
* Arterial hypertension (SBP < 160 mmHg and DBP < 100 mmHg)
* Patients, who tolerate ACEi treatment

Exclusion Criteria:

* Cholestasis, severe hepatic insufficiency
* Allergy to telmisartan
* Gravidity or lactation

Exclusion criteria for the arm of patient treated by ACEi:

* Cholestasis, severe hepatic insufficiency
* Allergy to ACEi
* Gravidity or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Any patient with a diagnosis of arterial hypertension, who do not tolerated ACE inhibitor treatment treated by the drug PRITOR
  * Exclusion criteria for the patients treated by the drug PRITOR must be read in conjunction with the local product information
Sampling Method: Non-Probability Sample
Enrollment: 3114 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy and safety of telmisartan in patients with arterial hypertension, who do not tolerate ACEI treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Many Locations, Romania
- Many Location, Slovakia